CLINICAL TRIAL: NCT05923970
Title: Is a Third Dose of Measles-mumps-rubella-(Varicella) Vaccine (MMR(V)) Vaccine Beneficial for the Adult Population in Alberta?
Brief Title: Is a Third Dose of MMRV Vaccine Beneficial for the Adult Population in Alberta?
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RES00059887
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Vaccination Failure; Vaccine Response Impaired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and isolated cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with low rubella antibodies: Women with rubella antibodies <10 IU/mL
  Interventions: Diagnostic Test: Serology for antibody levels - Baseline; Diagnostic Test: Serology to assess cell mediated immune (CMI) response - Baseline; Diagnostic Test: Serology for antibody levels - Post third dose of MMR vaccine; Diagnostic Test: Serology to assess CMI - Post third dose of MMR vaccine
- Women with high rubella antibodies: Women with rubella antibodies ≥10 IU/mL
  Interventions: Diagnostic Test: Serology for antibody levels - Baseline; Diagnostic Test: Serology to assess cell mediated immune (CMI) response - Baseline

INTERVENTIONS:
Diagnostic Test: Serology for antibody levels - Baseline — Measurement of rubella IgG antibody levels at baseline
Diagnostic Test: Serology to assess cell mediated immune (CMI) response - Baseline — Assessment of cell mediated immune (CMI) response to measles, mumps, rubella, and varicella at baseline.
Diagnostic Test: Serology for antibody levels - Post third dose of MMR vaccine — Measurement of rubella IgG antibody levels post third dose of MMR vaccine
  Groups: Women with low rubella antibodies
Diagnostic Test: Serology to assess CMI - Post third dose of MMR vaccine — Assessment of cell mediated response (CMI) to measles, mumps, rubella, and varicella post third dose of MMR vaccine.
  Groups: Women with low rubella antibodies

SUMMARY:
The current recommendation for a full course of measles-mumps-rubella-(varicella) vaccine (MMR(V)) is two doses. The problem is, many individuals within the vaccinated cohort show antibody levels that are below the level considered to be protective, even after two doses of vaccine. Because of these waning antibody levels, it is currently unknown whether highly vaccinated populations are protected from infection against measles, mumps, rubella, or varicella should they be exposed to any of these viruses. The uncertainty of a woman's immune status is partly due to the type of testing that is used to indicate protection. While immunity to viral infection requires both a humoral and a cell mediated immune (CMI) response, only humoral (antibody) responses are measured routinely in the laboratory. This study will examine CMI responses and the role of a third dose of vaccine for previously vaccinated women whose antibody levels are below the cut off. This study will not administer vaccine, but rather will include women who have received a third dose of vaccination through routine health care follow up in the study cohort.

DETAILED DESCRIPTION:
In highly vaccinated populations, the level of antibody produced against vaccine-preventable diseases has been waning overtime. Many low prevalence countries, including Canada, Israel, Australia, and Finland have reported decreases in the level of IgG for measles, mumps, rubella, and varicella often to below the level that is considered to be protective. These data have questioned the true level of protection in our populations. It is currently unclear if a vaccinated individual with low antibody levels, who was exposed to a vaccine preventable infection, would mount an effective immune response, or if they would develop infection. Susceptibility to infection is particularly concerning for prenatal populations, where exposure to rubella or varicella during pregnancy can result in congenital infection.

Rubella and varicella infection are considered mild, self-limiting illnesses when they affect young healthy children, however fetal infection during the first 16-20 weeks of gestation can result in development of congenital rubella syndrome (CRS), or congenital varicella syndrome (CVS). CRS is associated with severe long-term sequelae including microphthalmia, chorioretinitis, deafness, limb aplasia, and cognitive impairments such as microcephaly, while CVS is associated with skin lesions, neurological defects, limb hypoplasia, and can cause up to 20% fetal mortality. In endemic countries, CRS and CVS continue to be reported at high levels. Worldwide, approximately 100,000 CRS cases are estimated per year, while global estimates are not known for CVS, incidence rates of 1.6-4.3/1,000 were reported in the 1990's in the US. Prevention of these congenital conditions is therefore the primary goal of prenatal programs worldwide.

The standard laboratory method to determine if an individual has protective immunity against rubella and varicella infection is to test for circulating antibodies specific to rubella or varicella. Individuals with immunoglobulin G (IgG) antibody levels that are above the assay cut off (>10 IU/ml for rubella and positive for varicella) are considered protected from infection, while individuals with IgG levels that are below the cut off are considered susceptible to infection. Recently, our group has examined the longevity of anti-rubella and anti-varicella IgG levels in pre- and post-vaccination cohorts in the Alberta prenatal population. Following introduction of universal childhood vaccination programs, the level of IgG has decreased relative to age. For rubella, individuals who were born in or after 1981, and for varicella, individuals who were <20 years of age, have significantly lower rubella or varicella IgG levels respectively than those who were born prior to universal childhood vaccination programs (and whose immunity is derived by natural infection). Decreasing antibody levels for rubella, measles, and mumps have also been described in other vaccinated populations, suggesting that waning immunity is specific to populations where endemic transmission has been eliminated, or significantly reduced.

It is difficult to determine whether women whose antibody levels are detectable, but below the protective cut off, would mount a protective immune response upon challenge of viable virus. Disconcertingly, 30% of women undergoing prenatal screening in Alberta with low antibody levels against rubella previously received a full vaccine course (2 doses of a rubella containing vaccine). It is currently unknown whether these vaccinated women would mount an effective immune response, without additional vaccination, or if their infants would be at risk for CRS.

The uncertainty of a woman's immune status is partly due to the type of testing that is used to indicate protection. While immunity to viral infection requires both a humoral and a cell mediated immune (CMI) response, only humoral (antibody) responses are measured routinely in the laboratory.

The live-attenuated measles/mumps/rubella/varicella viruses used in vaccine closely mimic interactions that would be observed between the host and a wild type virus. The attenuated vaccine virus is known to replicate within host cells, similar to wild type virus, and can be detected in the blood of volunteers following vaccination. T cell responses have been shown to be long-lived following vaccination, for example T cell proliferation was observed following rubella-specific peptide stimulation 14-16 years after a single dose of vaccine. Likewise, in children who were vaccinated with live attenuated measles vaccine, only 1.90/100,000 where infected during a measles outbreak in the population 10 years later, while 17.84/100,000 children who received a killed vaccine (which would not effectively stimulate the CMI response), were infected during the same measles outbreak. In the context of herd immunity, low (but detectable) antibody levels may be sufficient to provide immunity to rubella infection, however no correlation between antibody levels and CMI has been performed for large, vaccinated populations.

This study will examine CMI responses and the role of a third dose of vaccine for previously vaccinated women whose antibody levels are below the cut off. This study will not administer vaccine, but rather will include women who have received a third dose of vaccination through routine health care follow up in the study cohort. Rubella antibody levels will be used to separate women into high and low antibody groups. Measles, mumps, rubella, and varicella IgG levels and CMI responses will be measured pre- and post-third vaccine dose to determine the benefits of third dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant and have undergone routine prenatal screening for rubella antibodies.

Exclusion Criteria:

* Women younger than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: All women who undergo routine prenatal screening for rubella antibodies in Alberta are eligible to participate. The study population will include 100 women with rubella antibodies below 10 IU/ml, and 100 women with antibody levels >=10 IU/ml.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in rubella antibody level. | Change in level from baseline to 12 months.
  Change in immunoglobulin G (IgG) antibody level from baseline to post-receipt of a third dose of MMR vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No